CLINICAL TRIAL: NCT05746780
Title: Clinical Value and Prognostic Impact of Bilateral Elective Neck Dissection in Salvage Total Laryngectomy of cN0 Cases
Brief Title: Bilateral Elective Neck Dissection in Salvage Total Laryngectomy
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Galli Jacopo, Professor, head of dept. of Otorinolaringology, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3364
Record Dates: First submitted 2023-02-02; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Neck Cancer; Larynx; Larynx Cancer; Neck
Keywords: neck dissection; SALVAGE TOTAL LARYNGECTOMY
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Diseases; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Elective bilateral neck dissection in cN0 patients — Radical modified type 3 selective bilaterale elective neck dissection

SUMMARY:
The aim of this study is to evaluate the role of elective bilateral neck dissection in patients with clinically negative lymph nodes (cN0) who underwent salvage total laryngectomy, by estimating the prevalence of histologically positive occult lymph nodes (pN+). Secondary objective will be the assessment of complication rate and the evaluation of 5-year Overall Survival (OS) and 5-year Disease-Specific Survival (DSS) in these patients.

ELIGIBILITY:
Inclusion criteria

-patients affected by recurrent laryngeal cancer after primary treatment failure (surgery or radiotherapy or chemoradiotherapy), with no clinical or radiological evidence of lymph node metastasis in the neck (cN0),who underwent salvage total laryngectomy and concomitant bilateral elective neck dissection (levels II, III, IV and VI).

Exclusion Criteria:

* patients who received other salvage laryngeal resection such as open partial horizontal laryngectomy, endoscopic partial laryngectomy, or who did not undergo bilateral selective neck dissection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient affected by recurrent laryngeal cancer, after failure of primary radiotherapy or conservative surgery, with clinically negative neck (cN0) and treated with salvage total laryngectomy and concomitant elective selective bilateral neck dissection (levels II-IV + VI).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Occult lymph node metastasis | At the time of salvage surgery
  Incidence rate of occult lymph node metastasislaryngectomy with clinically negative lymph nodes (cN0), estimating the prevalence of histologically positive lymph nodes (pN+) and predictive factors for cervical lymph nodes metastasis

SECONDARY OUTCOMES:
Complications of bilateral neck dissection during hospitalization | Up to 15 days from salvage surgery
  Complications of bilateral neck dissection during hospitalization
Overall survival | 5 year
  Survival of the patient from any disease
Disease specific survival | 5 years
  Survival of the patient from laryngeal disease

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Settimi, Roma, Italy

IPD SHARING:
Plan to Share IPD: No